CLINICAL TRIAL: NCT00083954
Title: A Confirmatory Multicenter, Double-blind, Randomized, Placebo Controlled Study of the Use of Quetiapine Fumarate (SEROQUEL) in the Treatment of Patients With Bipolar Depression
Brief Title: Controlled Study of the Use of Quetiapine Fumarate in the Treatment of Patients With Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D1447C00135
Record Dates: First submitted 2004-06-03; First posted 2004-06-07 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate

SUMMARY:
The purpose of this study is to determine the efficacy of quetiapine compared to placebo in the treatment for a major depressive episode in patients with bipolar disorder after receiving treatment for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before enrollment and any study-specific procedures. Patients deemed incapable of providing written consent will not be enrolled in this study; outpatient status

Exclusion Criteria:

* More than 8 mood episodes in the past year from screen (visit 1);
* A current Axis I disorder other than bipolar disorder within 6 months of screening;
* patients with clinically significant abnormal laboratory findings in the investigator's judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530
Dates: Start 2004-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 8 in the Montgomery-Asberg Depression Rating Scale (MADRS) total score

SECONDARY OUTCOMES:
Evaluate the incidence of treatment-emergent mania compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (36):
- United States (36):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Cerritos, California
  - Research Site, Garden Grove, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, Orlando, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Boise, Idaho
  - Research Site, Oak Brook, Illinois
  - Research Site, Overbrook Terrace, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Clementon, New Jersey
  - Research Site, Moorestown, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington

REFERENCES:
- [Derived] Lydiard RB, Culpepper L, Schioler H, Gustafsson U, Paulsson B. Quetiapine monotherapy as treatment for anxiety symptoms in patients with bipolar depression: a pooled analysis of results from 2 double-blind, randomized, placebo-controlled studies. Prim Care Companion J Clin Psychiatry. 2009;11(5):215-25. doi: 10.4088/PCC.08m00659. PMID 19956459